CLINICAL TRIAL: NCT02124811
Title: A Pilot Study of Minocycline Augmentation to Clozapine in Individuals With Treatment Resistant Schizophrenia
Brief Title: Minocycline Augmentation to Clozapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert Cotes, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00071195
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Clozapine; Minocycline
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High CRP (Experimental): Subjects with a High Baseline CRP will receive Minocycline. During the first week, subjects will receive one 100 mg capsule daily. On weeks 2-12, the subject will receive two 100 mg capsules at bedtime. The blinded psychiatrist (blinded to CRP status) will be allowed to reduce the dose if the subject complains of any side effect. Pending tolerability, the subject will have 200 mg per day.
  Interventions: Drug: Minocycline
- Low CRP (Experimental): Subjects with a Low Baseline CRP will receive Minocycline. During the first week, subjects will receive one 100 mg capsule daily. On weeks 2-12, the subject will receive two 100 mg capsules at bedtime. The blinded psychiatrist (blinded to CRP status) will be allowed to reduce the dose if the subject complains of any side effect. Pending tolerability, the subject will have 200 mg per day.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline

SUMMARY:
The proposed pilot study will compare minocycline augmentation with clozapine in individuals with high vs low inflammation as measured by CRP. Investigators hypothesize that minocycline will be well tolerated and will result in an improvement in the symptoms of schizophrenia, cognition, as well as improve the quality of life for patients preferentially in patients with high CRPs. Investigators plan to use a variety of different scales to measure improvement in the varying symptoms of schizophrenia as well as cognitive function, which will be administered to patients at three week intervals for a total study time of twelve weeks. Investigators hypothesize that minocycline could prove to be an effective, well tolerated, and inexpensive medication for treatment resistant patients with schizophrenia whom have particular difficulties with social interactions, obtaining and maintaining employment, and overall quality of life. Furthermore, investigators hypothesize that the data obtained in this study will contribute to the ongoing exploration of the role of inflammation in the brain of patients with schizophrenia and help understand and target the role of various inflammatory markers in the pathophysiology and treatment of treatment resistant schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a major mental illness characterized by a variety of different symptoms including hallucinations, paranoia, difficulties with formulating and expressing thoughts, feelings similar to depression, and problems with cognitive processes. Individuals with schizophrenia are usually treated with a class of medications called anti-psychotics, which typically help alleviate some of the symptoms of the disorder. In general, anti-psychotic medications do not completely cure the disorder, and many patients are left with some degree of ongoing symptoms. Furthermore, it is estimated that 20-30% of individuals with schizophrenia are considered treatment refractory or resistant and do not respond to anti-psychotic medications. The Food and Drug Administration has approved one antipsychotic medication for use in patients who are considered to have treatment resistant schizophrenia (TRS). This medication, clozapine, has been shown to be beneficial for patients with TRS, though as many as 40-70% of patients fail to respond or are partially responsive to treatment with clozapine. In an extensive search of the medical and psychiatric literature, the study team has been impressed by the potential of minocycline, a tetracycline antibiotic, as an adjunctive therapy in patients with schizophrenia based on its reported neuroprotective and anti-inflammatory effects. It is a fairly inexpensive drug, well tolerated, and two randomized clinical trials have demonstrated favorable results in early-phase schizophrenia. Only one case series with two patients has investigated minocycline in patients with schizophrenia on clozapine. Minocycline is also an interesting medication for augmentation with clozapine, as investigators are interested in previous findings of increased inflammation in the brains of patients with schizophrenia and the potential role of inflammation in treatment resistant schizophrenia. Though there are many markers of increased inflammation in the brain, for this current study, investigators are interested in a general marker of inflammation called C-Reactive Protein (CRP). The study team hypothesizes that some patients may have increased levels of inflammation in the brain, as measured by the CRP level (drawn from peripheral blood), and that those patients with increased levels of CRP may respond better to augmentation with minocycline. The proposed pilot study will compare minocycline augmentation with clozapine in individuals with high vs low inflammation as measured by CRP. Investigators hypothesize that minocycline will be well tolerated and will result in an improvement in the symptoms of schizophrenia, cognition, as well as improve the quality of life for patients preferentially in patients with high CRPs. Investigators plan to use a variety of different scales to measure improvement in the varying symptoms of schizophrenia as well as cognitive function, which will be administered to patients at three week intervals for a total study time of twelve weeks. Investigators hypothesize that minocycline could prove to be an effective, well tolerated, and inexpensive medication for treatment resistant patients with schizophrenia whom have particular difficulties with social interactions, obtaining and maintaining employment, and overall quality of life. Furthermore, investigators hypothesize that the data obtained in this study will contribute to the ongoing exploration of the role of inflammation in the brain of patients with schizophrenia and help understand and target the role of various inflammatory markers in the pathophysiology and treatment of treatment resistant schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Mini International Neuropsychiatric Interview 6.0 diagnosis of schizophrenia or schizoaffective disorder
* Persistent symptoms of schizophrenia as measured by one of the following PANSS items: Total score ≥60, negative subscale ≥ 15, positive subscale ≥ 15, general psychopathology subscale ≥ 30
* Currently taking clozapine and the dose has been adjusted within 100 mg of study enrollment
* Currently taking clozapine for 3 months and documented clozapine level ≥ 350 ng/ml prior to study start
* No other psychotropic medication changes for one month prior to study enrollment
* No new psychosocial interventions for one month prior to study enrollment
* No prior experience on minocycline for greater than 1 week
* May be taking any other psychotropic, dermatologic, or gastrointestinal drugs

Exclusion Criteria:

* History of organic brain disease
* Diagnostic and Statistical Manual of Mental Disorders (DSM) IV-TR diagnosis of Mental Retardation or Dementia
* DSM-IV-TR diagnosis of Alcohol or Substance Dependence within the last six months (except nicotine)
* Pregnancy or lactation
* Known hypersensitivity to tetracyclines
* Current known infection
* Any known neurological disease or medical condition that could impact the measurement of the constructs being assessed
* Inpatient psychiatric hospitalization for worsening of psychiatric symptoms, OR worsening of symptoms requiring a new level of outpatient support, OR started on a new anti-inflammatory medication for greater than one week duration, OR addition of a new psychotropic medication for psychiatric symptom control
* A change in > 15% in PANSS score from the "Lead-In Visit" to the "M0 visit"

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Cotes, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Levkovitz Y, Mendlovich S, Riwkes S, Braw Y, Levkovitch-Verbin H, Gal G, Fennig S, Treves I, Kron S. A double-blind, randomized study of minocycline for the treatment of negative and cognitive symptoms in early-phase schizophrenia. J Clin Psychiatry. 2010 Feb;71(2):138-49. doi: 10.4088/JCP.08m04666yel. Epub 2009 Nov 3. PMID 19895780
- [Background] Chaudhry IB, Hallak J, Husain N, Minhas F, Stirling J, Richardson P, Dursun S, Dunn G, Deakin B. Minocycline benefits negative symptoms in early schizophrenia: a randomised double-blind placebo-controlled clinical trial in patients on standard treatment. J Psychopharmacol. 2012 Sep;26(9):1185-93. doi: 10.1177/0269881112444941. Epub 2012 Apr 23. PMID 22526685
- [Background] Kelly DL, Vyas G, Richardson CM, Koola M, McMahon RP, Buchanan RW, Wehring HJ. Adjunct minocycline to clozapine treated patients with persistent schizophrenia symptoms. Schizophr Res. 2011 Dec;133(1-3):257-8. doi: 10.1016/j.schres.2011.08.005. Epub 2011 Aug 26. No abstract available. PMID 21872445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2015 and November 2016 from the Persistent Symptoms: Treatment, Assessment and Recovery (PSTAR) Clinic at Grady Memorial Hospital in Atlanta, Georgia.
Pre-assignment Details: Eighteen individuals were screened and 8 of these did not meet eligibility criteria or were lost to follow up prior to beginning the study treatment, resulting in 10 participants who began treatment.
Groups:
- High CRP: Participants with treatment resistant schizophrenia and a high baseline C-reactive protein (CRP) level received minocycline augmentation with clozapine. CRP levels were measured by a high sensitivity CRP test (hs-CRP) and baseline values greater than 3 milligrams per liter (mg/L) of blood are considered high.
- Low CRP: Participants with treatment resistant schizophrenia and a low baseline C-reactive protein (CRP) level received minocycline augmentation with clozapine. CRP levels were measured by a high sensitivity CRP test (hs-CRP) and baseline values equal to or less than 3 milligrams per liter (mg/L) of blood are considered low.
Period: Overall Study
Arm/Group | High CRP | Low CRP
Started | 5 | 5
Completed | 2 | 3
Not Completed | 3 | 2
Not completed — Early termination | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High CRP | Low CRP | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Tumor Necrosis Factor (TNF) Alpha [Mean (Standard Deviation); unit: pg/ml] — Tumor necrosis factor (TNF) alpha is a cytokine associated with systemic inflammation and the normal range for TNF alpha is <5.6 picograms per milliliter (pg/ml).
  pg/ml | 6.07 (2.29) | 5.36 (2.88) | 5.71 (2.48)
Interleukin 1 (IL-1) beta [Mean (Standard Deviation); unit: pg/ml] — Interleukin 1 (IL-1) beta is a pro-inflammatory cytokine implicated in pain, inflammation and autoimmune conditions. The normal range for IL-1 beta is <3.9 pg/ml.
  pg/ml | 0.62 (0.20) | 0.73 (0.22) | 0.67 (0.21)
Interleukin 6 (IL-6) [Mean (Standard Deviation); unit: pg/ml] — Interleukin 6 (IL-6) is secreted by T cells and macrophages stimulating an immune response during infection and after trauma. The normal range for IL-6 is < 5 pg/ml.
  pg/ml | 3.12 (4.29) | 1.11 (0.21) | 2.12 (3.05)
Interleukin 10 (IL-10) [Mean (Standard Deviation); unit: pg/ml] — Interleukin 10 (IL-10) is a cytokine impacting immunoregulation and inflammation. The normal range for IL-10 is <2 pg/ml.
  pg/ml | 0.64 (0.56) | 0.23 (0.13) | 0.44 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Positive Subscale Score of the Positive and Negative Syndrome Scale (PANSS)
Description: Positive symptoms (representing unusual thought content) of schizophrenia/schizoaffective disorder were measured with the positive subscale of the Positive and Negative Syndrome Scale (PANSS). The PANSS is scored by the clinician-researcher after an interview with the patient and it is the most commonly used measure for assessing the symptoms of schizophrenia. Seven items measure the positive symptoms of delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The items are scored on a scale of 1 to 7 where 1 means the symptom is absent and 7 means the symptom is extreme. The total summed score for the positive subscale ranges between 7 and 49 where higher scores indicate more severe symptoms. A reduction in the score indicates an improvement in symptom severity.
Time Frame: Baseline, Week 12
Population: Participants who completed the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 22 (7.07) | 22.33 (1.53)
  Week 12 | 16 (5.66) | 20.33 (4.73)

2. Primary Outcome: Negative Subscale Score of the Positive and Negative Syndrome Scale (PANSS)
Description: Negative symptoms (representing a loss of normal functions) of schizophrenia/schizoaffective disorder were measured with the negative subscale of the Positive and Negative Syndrome Scale (PANSS). The PANSS is scored by the clinician-researcher after an interview with the patient and it is the most commonly used measure for assessing the symptoms of schizophrenia. Seven items measure the negative symptoms of blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity & flow of conversation, and stereotyped thinking. The items are scored on a scale of 1 to 7 where 1 means the symptom is absent and 7 means the symptom is extreme. The total summed score for the negative subscale ranges between 7 and 49 where higher scores indicate more severe symptoms. A reduction in the score indicates an improvement in symptom severity.
Time Frame: Baseline, Week 12
Population: Participants who completed the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 17 (12.73) | 22.67 (5.77)
  Week 12 | 16.5 (3.54) | 22.33 (2.08)

3. Primary Outcome: Brief Assessment of Cognition in Schizophrenia (BACS) Score
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is an instrument that assesses the aspects of cognition found to be most impaired and most strongly correlated with outcomes in patients with schizophrenia (verbal memory, working memory, motor speed, verbal fluency, attention and processing speed, and executive function). BACS takes less than 35 minutes to complete and was administered on an electronic tablet for this study. The composite score is a T-score that averages the standardized scale scores of each of the six tests. The composite T-score has a mean of 50 and a standard deviation of 10. Scores below 50 indicate lower than average cognition while scores above 50 indicate higher than average cognition. A prior study found that the BACS mean composite score for schizophrenia patients was 25.96 while healthy controls had a mean score of 47.00.
Time Frame: Baseline, Week 12
Population: This analysis includes participants who completed the study and who completed the BACS. One participant in the high CRP did not complete this test at either time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 1 | 3
units on a scale
  Baseline | 36 (0) | 31.33 (16.29)
  Week 12 | 42 (0) | 28 (13.00)

4. Primary Outcome: General Psychopathology Score of the Positive and Negative Syndrome Scale (PANSS)
Description: General symptoms of schizophrenia/schizoaffective disorder were measured using the general psychopathology subscale of the Positive and Negative Syndrome Scale (PANSS). The PANSS is scored by the clinician-researcher after an interview with the patient and it is the most commonly used measure for assessing the symptoms of schizophrenia. Sixteen items measure general psychopathology symptoms of somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance. Items are scored on a scale of 1 to 7 where 1 means the symptom is absent and 7 means the symptom is extreme. Total scores for this subscale can range from 16 to 112 where higher scores indicate more severe symptoms. A reduction in the score indicates an improvement in symptom severity.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 1 | 3
units on a scale
  Baseline | 33 (0.0) | 36 (7.55)
  Week 12 | 27 (0.0) | 37 (9.17)

5. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Score
Description: Perceived quality of life and general well being was assessed using the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). The Q-LES-Q-SF is a 16-item questionnaire asking participants to rate how satisfied they have been with heath related qualities on a 5-point scale where 1 = very poor and 5 = very good. Raw scores of the Q-LES-Q-SF range from 14 to 70 and higher scores indicate higher life enjoyment and satisfaction.
Time Frame: Baseline, Week 12
Population: Participants who completed the study are included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 47.5 (3.54) | 64 (14)
  Week 12 | 53.5 (10.61) | 65.67 (15.63)

6. Secondary Outcome: Global Assessment of Functioning (GAF) Score
Description: Social, occupational, and psychological functioning was to be assessed using the Global Assessment of Functioning (GAF) in the initial study protocol.
Time Frame: Baseline, Week 12
Population: A protocol amendment removed the GAF outcome measure as this information was determined to be non-essential. To reduce participant burden, data were not collected for this outcome measure.
Arm/Group | High CRP | Low CRP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time when participants begin taking the study medication until completion of study participation (after participants had taken the study medication for 12 weeks).
Description: Adverse Events and side effects were asked about using a Side Effect Checklist, which asks about common side effects of clozapine and minocycline and allow for an open ended question to capture any unanticipated adverse events.
Arm/Group | High CRP | Low CRP
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High CRP (N=5) | Low CRP (N=5)
Hospitalization due to ischemic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inpatient psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High CRP (N=5) | Low CRP (N=5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) — resolved by reducing blood pressure medications

LIMITATIONS AND CAVEATS:
The small sample size limits the conclusions that can be drawn from the data collected in this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes